CLINICAL TRIAL: NCT00000780
Title: A "Pre-Enrollment" Protocol for HIV-Infected Adolescents
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 220
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Adolescent Behavior
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Adolescent Behavior

SUMMARY:
PRIMARY: To identify, characterize, and co-enroll HIV-infected adolescents into existing and future ACTG (or other NIH-sponsored) HIV treatment protocols through the systematic and recurrent assessment of eligibility. To assess the ability of adolescents enrolled in ACTG 220 to adhere to ACTG (or other NIH-sponsored) HIV treatment protocols; and to define factors that influence the adolescent's ability to enter or adhere to study protocols.

SECONDARY: To describe the nature, stage, and progression of HIV infection in adolescents.

Little is known about HIV-infected adolescents as a group and, as a result, small numbers of them are currently enrolled in ACTG drug studies. Creative approaches are needed to encourage enrollment of HIV-infected adolescents whose socio-demographic profile has made access to NIH-sponsored research unlikely.

DETAILED DESCRIPTION:
Little is known about HIV-infected adolescents as a group and, as a result, small numbers of them are currently enrolled in ACTG drug studies. Creative approaches are needed to encourage enrollment of HIV-infected adolescents whose socio-demographic profile has made access to NIH-sponsored research unlikely.

At entry and at every subsequent visit, participants are systematically evaluated for eligibility and willingness to enter ACTG (or other NIH-sponsored) HIV treatment protocols from a menu developed and updated by the Pediatric Adolescent Working Group of the ACTG. A survey of participant attitudes, behaviors, and beliefs is administered and updated semiannually. Participants attend clinic visits every 3 months and are followed for a minimum of 6 months, until the end of the study. They receive periodic physical exams, STD and gynecologic or genitourinary evaluations, HIV symptom assessment and related diagnoses, TB evaluation, and laboratory tests (hematology and immunology).

ELIGIBILITY:
Inclusion Criteria

Participants must meet the following criteria:

* HIV infection.
* NOT currently enrolled in an ACTG treatment protocol.

Exclusion Criteria

Co-existing Condition:

Participants with the following condition are excluded:

* No legal provision for consent to participate in clinical research can be determined.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Overall Officials: D'Angelo LJ, Study Chair; Futterman D, Study Chair; Abdalian S, Study Chair
Locations (51):
- United States (48):
  - Univ of Alabama at Birmingham Schl of Med / Pediatrics, Birmingham, Alabama
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Children's Hosp of Los Angeles, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - George Washington Univ / Hershey Med Ctr, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Tulane Med Ctr Hosp, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Worcester Memorial Hosp / Med Ctr of Cntrl MA-Memorial, Worcester, Massachusetts
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - King's County Hosp Ctr / Pediatrics, Brooklyn, New York
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Children's Hosp Pact Prog / Children's Hosp of Buffalo, Buffalo, New York
  - Schneider Children's Hosp, New Hyde Park, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Montefiore Med Ctr Adolescent AIDS Program, The Bronx, New York
  - Westchester Hosp, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Cincinnati Children's Hosp / Univ Hosp, Cincinnati, Ohio
  - Univ of Cincinnati, Cincinnati, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - West Central Ohio Hemophilia Ctr / Children's Med Ctr, Dayton, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Univ Texas Health Science Ctr / Univ Texas Med School, Houston, Texas
  - Great Lakes Hemophilia Foundation, Wauwatosa, Wisconsin
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Fry LJ, Fernandez RA. HIV prevention: factors that predict compliance with testing and counseling procedures. J Am Osteopath Assoc. 1994 Oct;94(10):825-30. PMID 7814276
- [Background] D'Angelo LJ, Lindsey J, Zimmer B, Culnane M, Futtermann D. Attempting to enhance the enrollment of adolescents into AIDS clinical trials: the design of ACTG Protocol 220. AIDS Patient Care STDS. 1998 Nov;12(11):853-9. doi: 10.1089/apc.1998.12.853. PMID 11362042
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891